CLINICAL TRIAL: NCT05524545
Title: A Phase 1, Open-label, Multicenter, Safety, Pharmacokinetic, Pharmacodynamic Study of ALX148 in Combination With Enfortumab Vedotin and/or Other Anticancer Therapies in Subjects With Urothelial Carcinoma (ASPEN-07)
Brief Title: A Study of Evorpacept (ALX148) With Enfortumab Vedotin for Subjects With Urothelial Carcinoma (ASPEN-07)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ALX Oncology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASPEN-07
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Bladder Cancer; Urothelial Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — ALX148; enfortumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Evorpacept (ALX148) + Enfortumab Vedotin (Experimental): Phase 1a Dose Escalation: Evorpacept (ALX148) infusions will be administered every two weeks.
  Enfortumab vedotin will be administered at 1.25 mg/kg IV on Days 1, 8, and 15 of each 28-day cycle.
  Interventions: Drug: Evorpacept; Drug: Enfortumab Vedotin

INTERVENTIONS:
Drug: Evorpacept — Fusion protein that blocks CD47-SIRPalpha pathway
  Other Names: ALX148
Drug: Enfortumab Vedotin — Nectin-4 directed antibody and microtubule inhibitor conjugate
  Other Names: PADCEV

SUMMARY:
AT148007 is a Phase 1, open-label, multicenter, safety, pharmacokinetic, pharmacodynamic study of ALX148 in combination with enfortumab vedotin and/or other anticancer therapies in subjects with urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, unresectable locally advanced or metastatic urothelial carcinoma.
2. Must have received prior treatment with an immune checkpoint inhibitor (CPI).
3. Subjects must have received prior treatment with platinum-containing chemotherapy.
4. Subjects must have had progression or recurrence of urothelial cancer.
5. Subjects must have measurable disease according to RECIST (Version 1.1).
6. Adequate bone marrow function.
7. Adequate renal function.
8. Adequate liver function.
9. Adequate Eastern Cooperative Oncology Group (ECOG) performance status.

Exclusion Criteria:

1. Preexisting sensory or motor neuropathy Grade ≥2.
2. Presence of symptomatic or uncontrolled central nervous system (CNS) metastases.
3. Prior treatment with enfortumab vedotin or other monomethylauristatin (MMAE)-based antibody-drug conjugate (ADCs)
4. Prior treatment with any anti-CD47 or anti-signal regulatory protein-α (SIRPα) agent.
5. Known active keratitis or corneal ulcerations. Subjects with superficial punctate keratitis are allowed if the disorder is being adequately treated.
6. History of uncontrolled diabetes mellitus within 3 months of the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
First Cycle Dose limiting toxicities (DLTs) | Up to 28 days
Adverse Events (AEs) as characterized by type, frequency, severity (as graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v. 5.0)), timing, seriousness, and relationship to study therapy | Up to 24 months
Phase 1: Recommended Phase 2 Dose (RP2D) | Up to 15 months
  To identify the RP2D of ALX148 in combination with enfortumab vedotin

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusett's General, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - West Clinic, Germantown, Tennessee
  - UT Southwestern, Dallas, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington